CLINICAL TRIAL: NCT06013969
Title: Effisayil® REP:An Open-label, Multicenter, Single-arm, Post-marketing Trial (in Select Countries) to Evaluate Efficacy and Safety and the Impact of Immunogenicity on Efficacy, Safety, and Pharmacokinetics of Spesolimab i.v. in Treatment of Patients With Generalized Pustular Psoriasis (GPP) Presenting With a Recurrent Flare Following Their Initial GPP Flare Treatment With Spesolimab i.v.
Brief Title: A Study to Test Whether Spesolimab Helps People With Generalized Pustular Psoriasis (GPP) Who Need Treatment for Repeated Flares
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0120; 2022-502128-38-00 (Registry Identifier: CTIS); U1111-1291-3088 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GPP Patients (Experimental): Generalized Pustular Psoriasis (GPP) patients with a recurrent flare following initial GPP flare treatment with intravenous (i.v.) spesolimab.
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab intravenous (i.v.) infusion
  Other Names: Spevigo®

SUMMARY:
This study is open to adults with a serious skin disease called generalized pustular psoriasis (GPP) who have repeated flares of GPP. The purpose of this study is to find out whether a medicine called spesolimab helps people with repeated flares of GPP.

Participants are given a single dose of spesolimab as an infusion into a vein on the first day of an outbreak of GPP. They may be given a second dose 1 week later if doctors think it is helpful. They are also treated for additional GPP flares.

During the time of the study, doctors regularly examine participants' skin for signs of GPP to see how well the treatment works and take blood samples. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) pustulation sub-score of 0 or 1 and a known and documented history of Generalized Pustular Psoriasis (GPP) (per European Rare And Severe Psoriasis Expert Network - ERASPEN - criteria), regardless of Interleukin 36 Receptor Antagonist (IL-36RN) gene mutation status or Patients with a GPP flare and a known and documented history of GPP (per ERASPEN criteria) regardless of IL-36RN gene mutation status.
* Patients must have a history of frequent GPP flares in the past
* Male or female patients, aged ≥18 years (if local legislation for age of consent differs, then local legislation will be followed) at screening
* Signed and dated written informed consent prior to admission to the trial in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to start of any screening procedures
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly

Exclusion Criteria:

* Drug-triggered Acute Generalized Exanthematous Pustulosis (AGEP)
* Patients with primary plaque psoriasis vulgaris without presence of pustules or with pustules that are restricted to psoriatic plaques
* Patients with primary erythrodermic psoriasis vulgaris
* Patients with SAPHO (Synovitis-acne-pustulosis-hyperostosis-osteitis) syndrome
* Immediate life-threatening flare of GPP or requiring intensive care treatment, according to the investigator's judgement. Life-threatening complications mainly include, but are not limited to, cardiovascular/cytokine driven shock, pulmonary distress syndrome, or acute renal failure
* Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold upper limit normal (ULN) elevation in Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin
* Presence of acute demyelinating neuropathy
* Treatment with any drug considered likely to interfere with the safe conduct of the trial, as assessed by the investigator
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Achievement of a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) pustulation sub-score of 0 indicating no visible pustules at Week 1 | Up to week 1

SECONDARY OUTCOMES:
Achievement of a GPPGA pustulation sub-score of 0 or 1, with a ≥2-point reduction from baseline at Week 1 | Up to week 1

CONTACTS AND LOCATIONS:
Locations (35):
- United States (2):
  - University of California Irvine, Irvine, California
  - Red River Research Partners, LLC, Fargo, North Dakota
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Brazil (2):
  - Hospital Universitario Evangelico Mackenzie, Curitiba
  - Faculdade de Medicina do ABC, Santo André
- China (3):
  - Southern Medical University Dermatology Hospital, Guangzhou
  - Shanghai Skin Disease Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
- France (2):
  - HOP Trousseau, Chambray-lès-Tours
  - HOP Saint-Louis, Paris
- Germany (2):
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum der Universität München AÖR, München
- India (2):
  - SP medical college and associated group of hospitals, Bikaner
  - Nkp Salve Institute of Medical Sciences and Lata Mangeshkar Hospital, Nagpur
- ASST degli Spedali Civili di Brescia, Brescia, Italy
- Malaysia (7):
  - Hospital Selayang, Batu Caves
  - Hospital Pulau Pinang-Pulau Pinang-21953, Georgetown Pulau Pinang
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya
  - Sunway Medical Centre, Selangor Darul Ehsan
- National University Hospital-Singapore-42005, Singapore, Singapore
- Nelson Mandela Academic Clinical Research Unit (NeMACRU), Mthatha, Eastern Cape, South Africa
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (2):
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhonchiangmai Hospital, Muang Chiang Mai
- Tunisia (2):
  - Hedi Chaker Hospital, Department of Dermatology, Sfax
  - Farhat Hached Hospital, Sousse

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing